CLINICAL TRIAL: NCT02872974
Title: Consequences of Maternal Gestational Diabetes on Offspring's Cardiovascular Health: MySweetHeart Cohort
Brief Title: Gestational Diabetes and Offspring's Cardiovascular Health: MySweetHeart Cohort
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Nicole Sekarski, Associate Professor, University of Lausanne Hospitals
Other Study IDs: 2016-00745-C
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Cardiovascular Diseases; Gestational Diabetes Mellitus
Keywords: Cardiovascular diseases; Gestational diabetes mellitus; Pediatrics; Fetal programming; Cohort study
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exposed: Offspring of woman with GDM
  Interventions: Other: GDM
- Not exposed: Offspring of woman without GDM

INTERVENTIONS:
Other: GDM — Exposure to GDM during fetal life
  Groups: Exposed

SUMMARY:
MySweetHeart Cohort is an observational study to assess the effect of gestational diabetes mellitus (GDM) on early life offspring's cardiovascular health.

The primary objective is to assess the effect of GDM on the surrogate markers of cardiovascular disease (CVD) at birth (left ventricular mass index and subclinical atherosclerosis). The secondary objective is to assess the effect of GDM on the cardiovascular structure and function during the fetal period and neonatal adverse cardiovascular risk factors.

The main hypothesis is that offspring of women with GDM have a larger LVMI and a larger cIMT at birth (primary outcomes) compared with offspring of women without GDM. Further, other hypotheses are that offspring of women with GDM have more foetal cardiovascular alterations and adverse neonatal cardio-metabolic risk factors (secondary outcomes) compared with offspring of women without GDM.

My SweetHeart Cohort is linked to MySweetHeart Trial, a randomized controlled trial assessing the effect of a multidimensional interdisciplinary lifestyle and psychosocial intervention to improve the cardio-metabolic and mental health of women with GDM and their offspring. The principal investigators of this trial are Prof Jardena Puder and Dr Antje Horsch from Lausanne University Hospital.

ELIGIBILITY:
Inclusion Criteria:

Women aged 18 yrs or older, with or without GDM at 24-32 weeks of gestation, and understanding French or English.

Exclusion Criteria:

Women on strict bed-rest, with pre-existing diabetes or known severe mental disorder

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will include the offspring of 100 women with GDM and of 100 women without GDM. They will be recruited at 24-32 wks of gestation and will be followed-up with their offspring until birth. Primary outcomes will be measured shortly (2-7 days) after birth. Secondary outcomes will be measured during the foetal period (30-34 wks of gestation), at birth, and shortly (2-4 days) after birth. A long-term follow-up of these children is planned.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Left ventricular mass index | At birth
Carotid intima-media thickness | At birth

SECONDARY OUTCOMES:
Fetal cardiovascular alterations | 30-34 wks of gestation (During fetal life)
Fetal left ventricular mass index | 30-34 wks of gestation (During fetal life)
Fetal liver volume | 30-34 wks of gestation (During fetal life)
Cardiovascular risk factors | At birth

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Sekarski, Prof, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Plan to share data has to be defined

REFERENCES:
- [Derived] Di Bernardo SC, Lava SAG, Epure AM, Younes SE, Chiolero A, Sekarski N; MySweetHeart Research Group. Consequences of gestational diabetes mellitus on neonatal cardiovascular health: MySweetHeart Cohort study. Pediatr Res. 2023 Jul;94(1):231-238. doi: 10.1038/s41390-022-02390-4. Epub 2022 Nov 28. PMID 36443400
- [Derived] Epure AM, Di Bernardo S, Mivelaz Y, Estoppey Younes S, Chiolero A, Sekarski N; MySweetHeart Research Group. Gestational diabetes mellitus and offspring's carotid intima-media thickness at birth: MySweetHeart Cohort study. BMJ Open. 2022 Jul 26;12(7):e061649. doi: 10.1136/bmjopen-2022-061649. PMID 35882452
- [Derived] Horsch A, Gilbert L, Lanzi S, Gross J, Kayser B, Vial Y, Simeoni U, Hans D, Berney A, Scholz U, Barakat R, Puder JJ; MySweetHeart Research Group. Improving cardiometabolic and mental health in women with gestational diabetes mellitus and their offspring: study protocol for MySweetHeart Trial, a randomised controlled trial. BMJ Open. 2018 Feb 27;8(2):e020462. doi: 10.1136/bmjopen-2017-020462. PMID 29487077
- [Derived] Di Bernardo S, Mivelaz Y, Epure AM, Vial Y, Simeoni U, Bovet P, Estoppey Younes S, Chiolero A, Sekarski N; MySweetHeart Research Group. Assessing the consequences of gestational diabetes mellitus on offspring's cardiovascular health: MySweetHeart Cohort study protocol, Switzerland. BMJ Open. 2017 Nov 14;7(11):e016972. doi: 10.1136/bmjopen-2017-016972. PMID 29138200